CLINICAL TRIAL: NCT03266874
Title: Prospective Multicenter Observational Evaluation of the Use of the G7 BiSpherical Acetabular Shell
Brief Title: G7 BiSpherical Acetabular Shell PMCF Study
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: H.CR.I.EU.16.26
Record Dates: First submitted 2017-08-24; First posted 2017-08-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Noninflammatory Degenerative Joint Disease; Avascular Necrosis; Correction of Functional Deformity; Non-Union Fracture; Femoral Neck Fractures; Trochanteric Fractures
Keywords: total hip arthroplasty
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Osteonecrosis; Fractures, Ununited; Femoral Neck Fractures; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- Patients who received the G7 BiSpherical Cup: Subject in need of a THA who met the inclusion/exclusion criteria and received the G7 BiSpherical cup.

SUMMARY:
The primary objective of this study is to obtain implant survivorship and clinical outcomes data for the commercially available G7 BiSpherical Acetabular Shell.

DETAILED DESCRIPTION:
The G7 BiSpherical Acetabular Shell belongs to the G7 multi-bearing platform. It was developed to provide an additional surgical option for patients in need of a total hip replacement. The aim of the G7 BiSpherical Acetabular Shell is to increase hip function while reducing pain.

This study is a multicenter, prospective, non-randomized, non-controlled post market surveillance study involving orthopedic surgeons skilled in hip arthroplasty procedures. A minimum of 4 and a maximum of 5 sites will be involved in this study. This number of clinical centers will permit assessment of consistency among a multitude of investigators. 140-175 implants will be included into the study. Each site will be allowed to enroll 35 patients. All potential study subjects will be required to participate in the Informed Consent Process.

The safety and performance of the G7 BiSpherical Acetabular Shell will be assessed as following: implant survivorship based on revision with removal of the study device; safety based on incidence and frequency of adverse events; and clinical efficacy measured by overall pain and function, quality of life data and radiographic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patient capable of understanding the surgeon's explanations and following his instructions, able and willing to participate in the follow-up program and who gave consent to take part in the study.
* Patient aged of 18 years or more whose skeleton reached bone maturity.
* Noninflammatory degenerative joint disease including osteoarthritis and avascular necrosis.
* Rheumatoid arthritis.
* Correction of functional deformity.
* Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques.
* Revision procedures where other treatment or devices have failed.

Inclusion criteria specific for patients receiving the G7 BiSpherical Shell with the G7 Freedom Constrained Liner:

* The Biomet G7 Freedom Constrained Liner is indicated for use as a component of a total hip prosthesis in primary and revision patients at high risk of dislocation due to a history of prior dislocation, bone loss, joint or soft tissue laxity, neuromuscular disease, or intraoperative instability, and for whom all other options to con-strained acetabular components have been considered.

Exclusion Criteria:

Absolute exclusion criteria include:

* Infection, sepsis, osteomyelitis.

Relative exclusion criteria include:

* Uncooperative patient or patient with neurologic disorders who is incapable of following directions.
* Osteoporosis.
* Metabolic disorders which may impair bone formation.
* Osteomalacia.
* Distant foci of infections which may spread to the implant site.
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram.
* Vascular insufficiency, muscular atrophy or neuromuscular disease.
* Patient unwilling or unable to give consent, or to comply with the follow-up program.
* Patient known to be pregnant or breastfeeding.
* Patient presenting any condition that would, in the judgment of the Investigator, place the patient at undue risk or interfere with the study.
* Patient institutionalized or known drug abuser or alcoholic or anyone who cannot understand what is required of them.
* Patient belonging to a vulnerable population.

Exclusion criteria specific for patients receiving the G7 BiSpherical Shell with the G7 Freedom Constrained Liner:

* Bone or musculature compromised by disease, infection, or prior implantation that cannot provide adequate support or fixation for the prosthesis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in need of a Total Hip Arthroplasty (primary or revision) which receive the G7 BiSperical Acetabular Shell and who meet all of the inclusion and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2017-12-10 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Implant survivorship is assessed counting the number of implant revisions | 10 years

SECONDARY OUTCOMES:
Clinical efficacy of the device is assessed using the Oxford Hip Score patient questionnaire | 10 years
Clinical efficacy of the device is assessed using the Harris Hip Score patient questionnaire | 10 years
Safety is assessed according to the number of complications which are collected via adverse event forms. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (5):
- Cabinet du Dr. Miazzolo, Perpignan, France
- Germany (2):
  - Orthopädische Chirurgie Müchen OCM, Munich, Bavaria
  - Herzogin Elisabeth Hospital, Braunschweig, Lower Saxony
- Reinier de Graaf Groep, Delft, Netherlands
- Orthoprax AG, Bern, Switzerland